CLINICAL TRIAL: NCT06097299
Title: A Phase 2, Randomized, Observer-blind Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1345, an mRNA Vaccine Targeting Respiratory Syncytial Virus, in Children 2 to <18 Years of Age at High Risk of Respiratory Syncytial Virus Disease
Brief Title: A Study of mRNA-1345, an mRNA Vaccine Targeting Respiratory Syncytial Virus, in Children 2 to <18 Years of Age at High Risk of Respiratory Syncytial Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1345-P202; 2024-000502-15 (EudraCT Number)
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Syncytial Virus
Keywords: Pediatric; mRNA-1345; RSV vaccine; Viral Diseases; Messenger RNA; Moderna
MeSH Terms: conditions — Virus Diseases | interventions — mRNA-1345 respiratory syncytial virus vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A and Part B: Cohort 1 (2 to <5 Years of Age) (Experimental): Part A: Participants 2 to <5 years of age will receive either a single intramuscular (IM) injection of mRNA-1345 or placebo on Day 1. Part B: Participants will have the option to be re-enrolled into a 6-month safety-follow up period.
  Interventions: Biological: mRNA-1345; Biological: Placebo
- Part A: Cohort 2 (5 to <18 Years of Age) (Experimental): Participants 5 to <18 years of age will receive a single IM injection of mRNA-1345 on Day 1.
  Interventions: Biological: mRNA-1345

INTERVENTIONS:
Biological: mRNA-1345 — Sterile liquid for injection
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Part A and Part B: Cohort 1 (2 to <5 Years of Age)

SUMMARY:
Part A: The purpose is to evaluate the safety, reactogenicity, and immunogenicity of mRNA-1345 in children aged 2 to <5 years (Cohort 1) and in children at high risk of respiratory syncytial virus (RSV) disease 5 to <18 years of age (Cohort 2) to inform the dose level selection for the next phase of development (Phase 3).

Part B: The purpose is to provide surveillance for RSV disease for the next RSV season (6 months after re-enrollment) and safety follow-up for Cohort 1 participants that were enrolled and dosed in Part A.

ELIGIBILITY:
Key Inclusion Criteria:

Part A Cohort 1:

* 2 to <5 years of age at Day 1.
* Healthy, or with stable chronic conditions increasing the risk of RSV disease, per the clinical judgment of the Investigator.

Cohort 2:

* 5 to <18 years of age at Day 1.
* Participants with stable chronic conditions increasing the risk of RSV disease.
* Female participants of child-bearing potential may be enrolled in the study, if the participant: 1) has a negative urine pregnancy test at Screening and on the day of injection (Day 1); 2) has practiced adequate contraception or has abstained from all activities that could lead to pregnancy for 28 days prior to Day 1; 3) has agreed to continue adequate contraception through 90 days following injection; and 4) is not currently breastfeeding.

Part B: Cohort 1 Re-enrollment

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Enrolled and dosed in Part A of Cohort 1; either reached EoS for Part A or were dosed and subsequently discontinued from study for various reasons. This includes participants who were lost to follow-up, if they can be re-engaged.
2. Participant's parent(s)/LAR(s) has provided written informed consent for participation in this study.

Key Exclusion Criteria (All Cohorts):

* Acutely ill or febrile (temperature ≥38.0°Celsius [100.4°Fahrenheit]) within 72 hours prior to or at the Screening Visit or Day 1.
* History of a diagnosis or condition that, in the judgment of the Investigator, may affect study assessment or compromise participant safety.
* Has received or plans to receive any licensed or authorized vaccine ≤14 days prior to the study vaccine injection (Day 1) or plans to receive a licensed or authorized vaccine within 14 days after the study vaccine injection.
* Receipt of any prior systemic immunosuppressants. Short courses (<7 days) of oral corticosteroids are allowed if completed at least 3 months prior to enrollment.
* Receipt of RSV monoclonal antibodies within 6 months prior to enrollment in the study.
* Participated in an interventional clinical study within 28 days (6 months for a study assessing a product unlicensed/unauthorized in this age group in country of residence at time of enrollment) prior to the day of enrollment or plans to do so while enrolled in this study.

Part B: Cohort 1 Re-enrollment

1. Participant is currently enrolled in another interventional clinical study.

Note: Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 346 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to 7 days postinjection
Part A: Number of Participants with Unsolicited Adverse Events (AEs) | Up to 28 days postinjection
Part A: Number of Participants With Medically Attended AEs (MAAEs) | Day 1 through end of study (EOS; Month 6)
Part A: Number of Participants With Adverse Events of Special Interest (AESIs) | Day 1 through EOS (Month 6)
Part A: Number of Participants With Serious Adverse Events (SAEs) | Day 1 through EOS (Month 6)
Part A: Number of Participants With AEs Leading to Discontinuation | Day 1 through EOS (Month 6)
Part B: Number of participants With Respiratory syncytial virus-Respiratory tract disease (RSV-RTD), Respiratory syncytial virus- Lower Respiratory tract disease (RSV-LRTD), Severe RSV-LRTD, Very Severe RSV-LRTD and RSV Hospitalization | Day 1 through EOS (Month 6)

SECONDARY OUTCOMES:
Part A: Geometric Mean Titer (GMT) of Serum RSV Neutralizing Antibody | Day 1, Day 29, and Month 6
Part A: Geometric Mean Concentration (GMC) of Serum RSV Prefusion F Binding Antibody | Day 1, Day 29, and Month 6
Part A: Geometric Mean Fold Rise (GMFR) of Postbaseline/Baseline Neutralizing Antibody Titers and Binding Antibody Concentrations | Baseline to Day 29 and Month 6
Part A: Number of Participants With Seroresponse in RSV Neutralizing Antibody | Baseline to Day 29 and Month 6
  Seroresponse is defined as a postinjection titer >4-fold-rise if Baseline is >lower limit of quantification (LLOQ) or >4 × LLOQ if Baseline titer is <LLOQ in RSV neutralizing antibody titers at Day 29 and Month 6.
Part B: Number of Participants With AESIs | Day 1 through EOS (Month 6)
Part B: Number of Participants With SAEs | Day 1 through EOS (Month 6)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (47):
  - Velocity Clinical Research, Phoenix, Phoenix, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - Velocity Clinical Research - Banning, Banning, California
  - ASCADA Research, LLC - Family Medicine, Fullerton, California
  - Ark Clinical Research, Long Beach, California
  - Peninsula Research Associates (PRA), Rolling Hills Estates, California
  - D&H Doral Research Center, LLC, Doral, Florida
  - Kissimmee Clinical Research, Kissimmee, Florida
  - Accel Clinical, Largo, Florida
  - Med-Care Research, Miami, Florida
  - Accel Research Sites - Nona Pediatric Center, Orlando, Florida
  - SEC Clinical Research, Pensacola, Florida
  - D&H Tamarac Research Center, Tamarac, Florida
  - Javara, Inc., Fayetteville, Georgia
  - Velocity Clinical Research-Primary Pediatrics, Macon, Macon, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Alliance for Multispeciality Research, LLC, El Dorado, Kansas
  - Velocity Clinical Research-Kansas City, Overland Park, Kansas
  - Velocity Clinical Research - Lafayette, Lafayette, Louisiana
  - Velocity Clinical Research Metairie, Metairie, Louisiana
  - Great Lakes Research Institute, Southfield, Michigan
  - Pediatric & Adolescent Center, Southgate, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Velocity Clinical Research, Gulfport, Gulfport, Mississippi
  - Velocity Clinical Research- Albuquerque, Albuquerque, New Mexico
  - Velocity Clinical Research-Binghamton, Binghamton, New York
  - University of Rochester Medical Center (URMC) - Golisano Children's Hospital (GCH), Rochester, New York
  - Senders Pediatrics, South Euclid, Ohio
  - The Children's Hospital of Philadelphia - Pediatrics, Philadelphia, Pennsylvania
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Velocity Clinical Research - Providence, Providence, Rhode Island
  - Coastal Pediatric Research, Charleston, South Carolina
  - Tribe Clinical Research, Simpsonville, South Carolina
  - Elligo Clinical Research Center, Austin, Texas
  - REX Clinical Trials, LLC, Beaumont, Texas
  - Javara Inc (Conroe), Conroe, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - DM Clinical Research - CyFair, Houston, Texas
  - Village Pediatrics, Plano, Texas
  - Javara Inc/Texas Health Care, PLLC d/b/a/ Privia Medical Group-North Texas, Stephenville, Texas
  - Victoria Clinical Research Group, Victoria, Texas
  - Velocity Clinical Research - Salt Lake City, West Jordan, Utah
  - PI-Coor Clinical Research, LLC, Annandale, Virginia
  - Clinical Research Partners, Richmond, Virginia
  - National Clinical Research, Inc., Richmond, Virginia
- Panama (3):
  - CEVAXIN Chorrera, La Chorrera
  - CEVAXIN Avenida Mexico, Panama City
  - CEVAXIN 24 de Diciembre, Panama City